CLINICAL TRIAL: NCT04777435
Title: Therapeutic Orientation Test in Thrombotic Microangiopathy
Acronym: TOTEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL19_0075
Record Dates: First submitted 2021-02-19; First posted 2021-03-02 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Thrombotic Micro-angiopathy
Keywords: Nephrology; Complement; Thrombotic micro-angiopathy; Diagnostic; Haemolytic and Uraemic Syndrome
MeSH Terms: conditions — Disease; Hemolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Thrombotic micro-angiopathy (Experimental)
  Interventions: Diagnostic Test: Therapeutic orientation test for TMA

INTERVENTIONS:
Diagnostic Test: Therapeutic orientation test for TMA — Therapeutic orientation test for TMA performed on blood sample at inclusion, first visit at 1 month and last visit at 6 months.

SUMMARY:
Haemolytic and Uraemic Syndrome (HUS) is a serious disease requiring rapid diagnosis and management. The atypical HUS diagnosis has been greatly improved by anti-CS antibody (Eculizumab) wich block alternative complement pathway activation. To rise treatment success, Eculizumab introduction should be as early as possible. In some secondary HUS (infection, drugs…) complement is also involved as "second-hit".

To date, there is no tool to confirm complement involvement in a HUS at diagnosis stage. This study suggest to evaluate a therapeutic orientation test, in order to determine the complement implication in HUS diagnosis. The test evaluates the complement deposits on endothelial cell surface in vitro, compared to a normal human serum.

In order to determine the test performance, first the positive or negative results will be compared to the HUS clinical evolution, treated or not by the clinician with Eculizumab. Second, the test results will be compared to the presence of alternative complement pathway regulation abnormalities.

ELIGIBILITY:
Inclusion Criteria:

TMA with:

* mechanic haemolytic anemia, undetectable haptoglobin, LDH>1.5*LNS
* thrombopenia
* acute kidney injury TMA on native kidney or in post-transplantation.

Exclusion Criteria:

* DIVC patients
* plasma exchange during 1 month before sample collection
* treatment by Eculizumab before sample collection
* no consent
* not beneficiary of a social security
* pregnancy or breastfeeding
* patient Under guardianship

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-03 (Actual); Primary Completion 2026-10-03 (Estimated); Study Completion 2027-04-03 (Estimated)

PRIMARY OUTCOMES:
Therapeutic orientation test sensitivity | Through study completion, an average of 3 years.
  The proportion of patients testing positive among those receiving a relevant Eculizumab treatment ( TMA resolution with treatment or presence of abnormalities in alternative complement pathway.
Therapeutic orientation test specificity | Through study completion, an average of 3 years.
  The proportion of patients testing negative among patients who did not receive Eculizumab treatment.(TMA resolution without treatment or therapeutic failure with Eculizumab).

SECONDARY OUTCOMES:
Untreated test positive patients | Through study completion, an average of 3 years.
  The proportion of patients with positive test but untreated by Eculizumab, and who therefore could have benefited from treatment.

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU de Bordeaux, Bordeaux
  - Site Médipôle Cabestany, Cabestany
  - Centre Nephrocare Castelnau-le-Lez, Castelnau-le-Lez
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - APHM-Hôpital de la Conception, Marseille
  - Montpellier University Hospital, Montpellier
  - CHU de Nantes, Nantes
  - HPGN- Narbonne, Narbonne
  - CHU de Nice, Nice
  - CHU de Nîmes, Nîmes
  - APHP-Hôpital Tenon, Paris
  - Hôpital Paris Necker, Paris
  - CH de Perpignan, Perpignan
  - CHU de Poitiers, Poitiers
  - CHU de Rouen, Rouen
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHRU Tours, Tours